CLINICAL TRIAL: NCT02480777
Title: Expanded Access for Single Patient Treatment of Autologous Human Schwann Cells (ahSC) for Peripheral Nerve Repair
Status: No longer available | Type: Expanded Access
Sponsor: W. Dalton Dietrich (Other)
Collaborators: The Miami Project to Cure Paralysis (Other)
Responsible Party: Sponsor-Investigator, W. Dalton Dietrich, Professor of Neurosurgery, University of Miami
Organization: University of Miami (Other)
Other Study IDs: 20130722
Record Dates: First submitted 2015-06-21; First posted 2015-06-25 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Sciatic Nerve Injury

INTERVENTIONS:
Biological: Autologous Human Schwann cells — Schwann cells harvested from the sural nerve and debrided, injured sciatic nerve of the participant will be autologously transplanted along sural nerve autografts wrapped in a collagen matrix (Duragen).

SUMMARY:
The primary purpose of this research study is to determine the safety of injecting ones own Schwann cells as a supplement along with nerve autograft (eg sural nerve) a few weeks after a severe injury to the sciatic nerve has occurred.

DETAILED DESCRIPTION:
The secondary purpose of this research project is to evaluate whether transplanted Schwann cells can enhance recovery of sensory and motor function. Emergency expanded access for a single patient was granted, as the patient was an ideal candidate for sural nerve repair augmented by autologous Schwann cells which could be harvested either from a relatively small segment of sensory nerve or as in this case from local debridement of injured nerve at the epicenter of the nerve injury. The cells were expanded using cell culture techniques and placed along with the sural nerve grafts wrapped by an FDA approved collagen matrix (Duragen). This study is being conducted at the Jackson Memorial and the University of Miami health systems. As a research subject the patient will be in this study for a total of 5 years from the date receiving Schwann cell transplant augmentation of sural nerve autografts.

ELIGIBILITY:
- single patient with severe sciatic nerve injury enrolled under emergency request

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Allan Levi, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States